CLINICAL TRIAL: NCT03503448
Title: Clinical Trial Comparing 2 Techniques of Surgically Assisted Rapid Maxillary Expansion
Brief Title: Comparison of 2 Techniques of Surgically Assisted Rapid Maxillary Expansion
Acronym: SARME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Pedro Ernesto (Other)
Responsible Party: Principal Investigator, Pedro Andre Alves Pereira, DDS, Clinical Research, Hospital Universitario Pedro Ernesto
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69696317.0.0000.5259
Record Dates: First submitted 2018-04-01; First posted 2018-04-19 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Malocclusion; Maxillar Hypoplasia; Transverse Maxillary Deficiency
Keywords: surgically assisted rapid maxillary expansion; surgically assisted rapid palatal expansion; Malocclusion
MeSH Terms: conditions — Malocclusion; Retrognathia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- space between 11/21 (Other): Osteotomy between the maxillary central incisors
  Interventions: Procedure: Osteotomy between the maxillary central incisors
- space between 12/13 and 22/23 (Other): Osteotomy between the maxillary lateral incisors and canines
  Interventions: Procedure: Osteotomy between the maxillary lateral incisors and canines

INTERVENTIONS:
Procedure: Osteotomy between the maxillary central incisors — Surgically Assisted Rapid Maxillary Expansion with osteotomy between the central incisors.
  Arms: space between 11/21
Procedure: Osteotomy between the maxillary lateral incisors and canines — Surgically Assisted Rapid Maxillary Expansion with bilateral osteotomy between the lateral incisors and canines
  Arms: space between 12/13 and 22/23

SUMMARY:
This study evaluates 2 Techniques of Surgically Assisted Rapid Maxillary Expansion (SARME) in the treatment of maxillary transverse deficiency. Half of participants will undergo an osteotomy between the maxillary central incisors, while the other half will undergo an osteotomy between the maxillary lateral incisors and canines (bilateral osteotomies).

DETAILED DESCRIPTION:
Surgically Assisted Rapid Maxillary Expansion (SARME) can be performed by a osteotomy between the maxillary central incisors and by osteotomies between the maxillary lateral incisors and canines (bilateral).

Both techniques treat transverse maxillary hypoplasia, but they do so with different effects on esthetics, periodontium, teeth and bone expansion.

ELIGIBILITY:
Inclusion Criteria: patients with bilateral cross-bite and bilateral transverse maxillary deficiencies equal to or greater than 6 mm -

Exclusion Criteria: Patients with previous histories of maxillary surgery, congenital craniofacial malformations, unilateral transverse maxillary deficiencies and absence of teeth in the maxilla.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Bone expansion and dental inclination | 1-2 months post-expansion.
  Assessment of bone expansion and dental inclination through Cone Beam computed tomography (CBCT) images

SECONDARY OUTCOMES:
Patient´s perception | 2 months post-expansion.
  Patient´s cosmetic perception of his or her smile on a visual analogue scale (VAS) ranging from 0 to 10, where "0" represents total dissatisfaction and "10" represents total satisfaction with the postoperative smile.
Periodontal effects | 2 months post-expansion.
  Assessment of periodontal changes in the teeth adjacent to the segmentation, through periodontal probing
Surgery time | During surgery
  Time elapsed during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio G Ritto, PhD, Study Chair — Hospital Universitario Pedro Ernesto
Locations (1):
- Hospital Universitario Pedro Ernesto, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No
I plan to share the data on March 24, 2020 when I going to present my Master degrees' thesis. I tried to submit an article with the data. I'm waiting for a reply

REFERENCES:
- [Result] Landes CA, Laudemann K, Petruchin O, Mack MG, Kopp S, Ludwig B, Sader RA, Seitz O. Comparison of bipartite versus tripartite osteotomy for maxillary transversal expansion using 3-dimensional preoperative and postexpansion computed tomography data. J Oral Maxillofac Surg. 2009 Oct;67(10):2287-301. doi: 10.1016/j.joms.2009.04.069. PMID 19761925
- [Result] Betts NJ. Surgically Assisted Maxillary Expansion. Atlas Oral Maxillofac Surg Clin North Am. 2016 Mar;24(1):67-77. doi: 10.1016/j.cxom.2015.10.003. Epub 2015 Nov 24. No abstract available. PMID 26847514
- [Result] Camps-Pereperez I, Guijarro-Martinez R, Peiro-Guijarro MA, Hernandez-Alfaro F. The value of cone beam computed tomography imaging in surgically assisted rapid palatal expansion: a systematic review of the literature. Int J Oral Maxillofac Surg. 2017 Jul;46(7):827-838. doi: 10.1016/j.ijom.2017.01.017. Epub 2017 Mar 6. PMID 28279603